CLINICAL TRIAL: NCT06152146
Title: Randomized Controlled Trial of Low Intensity Shockwaves Therapy for the Treatment of Post-Radical Prostatectomy Erectile Dysfunction. SHARP-ED TRIAL
Brief Title: Clinical Trial of Low Intensity Shockwaves Therapy for Erectile Dysfunction Post-Radical Prostatectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study submission was discarded with the IRB and no longer moving forward
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Russell Saltzman, Regulatory Specialist, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20231090
Record Dates: First submitted 2023-10-10; First posted 2023-11-30 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SWT group (Active Comparator): Participants randomized to the treatment group will receive nine (9) shockwave sessions in total: one (1) shockwave session once per week for four (4) weeks, followed by one (1) shockwave session once per month (30±7 days) for the next five (5) months. 1,440 shocks of treatment energy will be applied in every session to each treated region (left and right corpora cavernosa and crura) for a total of 12,960 shocks. Participants will be in this group for up to 6 months.
  Interventions: Device: Shockwave Therapy
- SHAM group (Placebo Comparator): Participants randomized to the sham (control) group will have nine (9) sham therapy sessions in total: one (1) sham session once per week for four (4) weeks, followed by one (1) sham session once per month (30±7 days) for the next five (5) months. The shockwave machine will be set to deliver 1,440 shock treatments, but a barrier will be placed around the shockwave probe to ensure that no shockwaves are delivered. Participants will be in this group for up to 6 months.
  Interventions: Other: SHAM shockwave therapy

INTERVENTIONS:
Device: Shockwave Therapy — Each therapy session will last about 20 minutes, during which 1,440 shockwaves will be applied to the penis via the left and right crus (shaft near the base)
  Arms: SWT group
Other: SHAM shockwave therapy — Each therapy session, lasting about 20 minutes, will deliver 1440 SHAM shockwave therapy applied to the penis via the left and right crus (shaft near the base)
  Arms: SHAM group

SUMMARY:
Research study designed to learn about and compare Shockwave therapy (SWT) vs placebo (no shockwaves) treatment in men with moderate to severe erectile dysfunction (ED) after Radical Prostatectomy

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide informed consent.
2. Be male
3. Be ≥ 40 and ≤ 75 years of age (inclusive).
4. Undergo radical prostatectomy for prostate cancer (nerve sparing or non-nerve sparing without neoadjuvant chemotherapy or radiation therapy.)
5. Be at least six weeks post radical prostatectomy.
6. Be in a stable sexual relationship for over 3 months prior to enrollment.
7. Have testosterone level of 300-1000 ng/dL within 1 month prior to enrollment.
8. Have an HbA1c level ≤ 7% within 3 months prior to enrollment.
9. Have undetectable PSA value at the time of enrollment

Exclusion Criteria:

1. Be currently participating in a clinical trial or have recently received an investigational therapy within the past 30 days that may interfere with the results of this study.
2. Be under judicial protection (prison or custody).
3. Be an adult under guardianship.
4. Refuse to sign the informed consent.
5. Have evidence of venous leak prior to surgery or use of PDE5i prior to surgery
6. Have past radiation therapy of the pelvic region or hormonal therapy with androgen deprivation within 12 months prior to enrollment.
7. Be recovering from any cancer within 12 months prior to enrollment (other than prostate cancer)
8. Have Neurological disease such as Alzheimer's or Parkinson's disease which affects erectile function (at the discretion of the investigator).
9. Have a Psychiatric diagnosis or medications such as antidepressants, anxiolytic, antipsychotic that affects erectile function or any other medications (at the discretion of the investigator).
10. Have an anatomical malformation of the penis, including Peyronie's disease.
11. Have testosterone level <300 or >1000 ng/dL within 1 month prior to enrollment.
12. Be using blood thinners with international normalized ratio (INR) to be > 3.
13. Have received shockwave therapy for at least 6 months before enrollment.
14. Have detectable PSA value after the radical prostatectomy.
15. Require radiation therapy after radical prostatectomy.
16. Require hormonal therapy after radical prostatectomy.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-08 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in number of participants reporting on Penetrative Intercourse | Baseline to 6 months and Baseline to 12 months.
  Number of participants reporting the ability to have penetrative intercourse with or without PDE5i but without the use of intracavernosal injections was chosen as the primary clinical efficacy assessment tool in this study.

SECONDARY OUTCOMES:
Change in Penile blood flow (Penile Duplex Ultrasound) measured in centimeters per second (cm/sec) | Baseline to 12 months.
  Penile Blood Flow will be reported as Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV), both assessed in cm/sec, via Penile Doppler ultrasonography
Change in IIEF-EF Scores | Baseline to 6 months and Baseline to 12 months.
  The International Index of Erectile Function - Erectile Function ( domain score is a patient questionnaire (six questions) used to measure various aspects of erectile performance and assess disease severity in efficacy trials concerning ED. The International Index of Erectile Function - Erectile Function has a minimum score of 0 and max of 30, higher scores mean a better outcome.
Change in SEP- Sexual Encounter Profile: Questions 2 and 3 | Baseline to 6 months and Baseline to 12 months.
  The Sexual Encounter Profile (SEP) is a log diary completed after each sexual attempt, providing information as to whether the erection was hard enough to penetrate (SEP 2), or whether it was maintained for completion (SEP 3). Mixed effect linear regression will be used to model post randomization repeated measurements of continuous outcomes. From the results of the model, the mean difference between groups at each time point will be estimated along with a 95% confidence interval.
Change in GAQ- Global Assessment Questions | Baseline to 6 months and Baseline to 12 months.
  The Global Assessment Questions is a measure of perceived improvements in erectile function and sexual ability. It also evaluate improvements in erectile function and ability to engage in sexual activity. The Scoring: GAQ is comprised of two 'yes or no' questions with a total score ranging from 0-2. Categorical data can be obtained from this measure
Change in EHS- Erection Hardness Score | Baseline to 6 months and Baseline to 12 months.
  The Erection Hardness Score (EHS) is a single-item, patient-reported outcome (PRO) for scoring erection hardness. The EHS consists of a single question and the responses are scored from 0-4 with higher scored indicating more erection hardness.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — University of Miami
Locations (1):
- Desai Sethi Urology Institute - University of Miami, Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No